CLINICAL TRIAL: NCT07262710
Title: Association of Angiotensin-Converting Enzyme Inhibitors and Angiotensin Receptor Blockers With Post-Stroke Pneumonia: A Real-World Retrospective Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xiaonong Fan, Chief physician, First Teaching Hospital of Tianjin University of Traditional Chinese Medicine
Other Study IDs: XFan
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Post-stroke Pneumonia
Keywords: post-stroke pneumonia; angiotensin converting enzyme inhibitors; angiotensin receptor blockers
MeSH Terms: interventions — Angiotensin-Converting Enzyme Inhibitors; Calcium Channel Blockers; Angiotensin Receptor Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ACEI-exposed group: Newly Initiated ACEI
  Interventions: Drug: angiotensin converting enzyme inhibitors
- ARB-exposed group: Newly Initiated ARB
  Interventions: Drug: Angiotensin Receptor Blockers
- CCB-exposed group1: Newly Initiated CCB
  Interventions: Drug: Calcium Channel Blockers
- CCB-exposed group2: Newly Initiated CCB
  Interventions: Drug: Calcium Channel Blockers

INTERVENTIONS:
Drug: angiotensin converting enzyme inhibitors — The Angiotensin-Converting Enzyme Inhibitors (ACEIs) in this study included Captopril, Enalapril, Lisinopril, Perindopril, Ramipril, Quinapril, Benazepril, Cilazapril, Fosinopril, Trandolapril, Spirapril, Delapril, Moexipril, Temocapril, Zofenopril, and Imidapril.
  Groups: ACEI-exposed group
Drug: Calcium Channel Blockers — The Calcium Channel Blockers (CCBs) evaluated as the active comparator in this study comprised a comprehensive list, including Amlodipine, Felodipine, Isradipine, Nicardipine, Nifedipine, Nimodipine, Nitrendipine, Lacidipine, Nilvadipine, Manidipine, Barnidipine, Lercanidipine, Cilnidipine, Benidipine, Clevidipine, Mibefradil, Verapamil, Gallopamil, Diltiazem, Fendiline, and Bepridil.
  Groups: CCB-exposed group1; CCB-exposed group2
Drug: Angiotensin Receptor Blockers — The Angiotensin Receptor Blockers (ARBs) included in this analysis were Losartan, Eprosartan, Valsartan, Irbesartan, Candesartan, Telmisartan, Olmesartan Medoxomil, Azilsartan Medoxomil, and Fimasartan.
  Groups: ARB-exposed group

SUMMARY:
The goal of this retrospective cohort study is to determine if Angiotensin-Converting Enzyme Inhibitors (ACEIs) and Angiotensin Receptor Blockers (ARBs) can lower the risk of post-stroke pneumonia. With an active comparator, new-user design, we selected new users of Calcium Channel Blockers (CCBs) as the reference group to compare against new users of ACEIs/ARBs.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of both stroke and hypertension, with the initial diagnosis dates for both conditions falling within the period from January 1, 2016, to December 31, 2024.Definition of Stroke: International Classification of Diseases, 10th Revision (ICD-10) codes I60-I64, or a primary diagnosis of stroke-related conditions in inpatient/outpatient medical records, including but not limited to: cerebral hemorrhage, hemorrhagic stroke, cerebral infarction, ischemic stroke, cerebral ischemia, brainstem infarction.Definition of Hypertension: ICD-10 code I10, or inpatient/outpatient medical records containing diagnostic names such as hypertension, benign hypertension, hypertensive crisis.
2. At least one prescription filled from any of the five major classes of antihypertensive medications: Angiotensin-Converting Enzyme Inhibitors (ACEI), Angiotensin II Receptor Blockers (ARB), Beta-blockers, Calcium Channel Blockers (CCB), or Diuretics. Furthermore, there must be no record of any ACEI, ARB, or CCB prescriptions within the 12 months immediately preceding the first ACEI, ARB, or CCB prescription.
3. Aage ≥18 years.

Exclusion Criteria:

1. Data anomalies or errors(such as an inaccurately recorded date of death).
2. Concurrent use of two or three drug classes among ACEI, ARB, and CCB at any time.
3. Any recorded diagnosis of pneumonia prior to the initiation of the first antihypertensive medication.Definition of Pneumonia: ICD-10 codes J12-J18 or J69, or inpatient/outpatient medical records containing diagnostic names such as pulmonary infection, pneumonia, lung infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosis of both stroke and hypertension, with the initial diagnosis dates for both conditions falling within the period from January 1, 2016, to December 31, 2024
Sampling Method: Probability Sample
Enrollment: 13656 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-19 (Estimated)

PRIMARY OUTCOMES:
Occurrence of post-stroke pneumonia | The follow-up end point was defined as the earliest occurrence of any of the following events: a diagnosis of pneumonia, death, the date of the last available medical record in the database, or the end of the study period (December 31, 2024).

IPD SHARING:
Plan to Share IPD: Undecided